CLINICAL TRIAL: NCT00305435
Title: An Open Label Phase 2 Study Evaluating the Safety of Starting Dose of AMG 531 in Thrombocytopenic Japanese Subjects With Immune (Idiopathic) Thrombocytopenic Purpura
Brief Title: Safety Study of AMG 531 in Japanese Subjects With ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050162
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Thrombocytopenia in Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Keywords: AMG 531, ITP, Phase 2, Japanese
MeSH Terms: conditions — Purpura, Thrombocytopenic; Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- romiplostim (AMG-531) (Experimental)
  Interventions: Drug: Romiplostim (AMG-531)

INTERVENTIONS:
Drug: Romiplostim (AMG-531) — Romiplostim (AMG-531)

SUMMARY:
The purpose of the study is to evaluate the efficacy of starting dose of AMG 531 as measured by platelet counts by cohort dose-escalation design.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy of starting dose of AMG 531 as measured by platelet counts by cohort dose-escalation design.

ELIGIBILITY:
Inclusion Criteria: - Japanese patients with diagnosis of ITP according to the diagnostic criteria proposed by Research Committee for Idiopathic Hematopoietic Disorders of the Ministry of health, labor and welfare Exclusion Criteria: - Documented diagnosis of arterial thrombosis in the previous year; history of venous thrombosis and receiving anticoagulation therapy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Incidence of all adverse events including evaluation of antibody status | 1 year

SECONDARY OUTCOMES:
Proportion of subjects who achieve a platelet response | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Shirasugi Y, Ando K, Hashino S, Nagasawa T, Kurata Y, Kishimoto Y, Iwato K, Ohtsu T, Berger DP. A phase II, open-label, sequential-cohort, dose-escalation study of romiplostim in Japanese patients with chronic immune thrombocytopenic purpura. Int J Hematol. 2009 Sep;90(2):157-165. doi: 10.1007/s12185-009-0361-y. Epub 2009 Jun 20. PMID 19543952
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_46_AMP-2_20050162.pdf
- See also: FDA-approved Drug Labeling — http://www.nplate.com/